CLINICAL TRIAL: NCT06811415
Title: Tempromandibular Joint Reconstruction Via Computer-Assisted Surgery Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Taha Ibrahim, Assistant professor, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #R-OS-10-24-3149
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Temporomandibular Joint
Keywords: 3D printed templates; computer-assisted surgical simulation; costochondral graft; temporomandibular joint

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual Tmj reconstruction with rib graft (Other): All patients were placed in preoperative occlusion in CASS. The planned rib was harvested in the standard manner through an inframammary incision. The length of the rib was equal to the prefabricated template as calculated in the cranial-maxillofacial 3D reconstruction, and comprised at most 5 mm of cartilage. The cartilage was trimmed and contoured to facilitate the setting of the cartilage side properly into the center of the TMJ fossa. A 4-hole titanium plate was fixed with four bicortical screws as previously planned
  Interventions: Procedure: virtual temporomandibular joint reconstruction with costochondral graft

INTERVENTIONS:
Procedure: virtual temporomandibular joint reconstruction with costochondral graft — All patients were placed in preoperative occlusion in CASS. The planned rib was harvested in the standard manner through an inframammary incision. The length of the rib was equal to the prefabricated template as calculated in the cranial-maxillofacial 3D reconstruction, and comprised at most 5 mm of cartilage. The cartilage was trimmed and contoured to facilitate the setting of the cartilage side properly into the center of the TMJ fossa. A 4-hole titanium plate was fixed with four bicortical screws as previously planned

SUMMARY:
This study was planned to evaluate the accuracy of virtual surgical planning and three-dimensional (3D) printed templates in reconstruction of temporomandibular joint (TMJ) with costochondral graft.

DETAILED DESCRIPTION:
Eight patients (15-45) years diagnosed with TMJ deformities were included. A composite skull model was obtained with data from computed tomography. A virtual surgical simulation was performed using Dolphin Imaging 11.7 Premium. Then, the virtual plan was transferred to the operative field using 3D (CAD-CAM) printed surgical template. These templates were designed by 3D printing using data from the virtual surgical simulation for optimum selection of the rib graft, accurate tailoring of chondral and costal graft and as an osteotomy guide.

The preoperative measurement including mouth opening, facial asymmetry and differences between the actual mandibular position and the virtual plan were analyzed

ELIGIBILITY:
Inclusion Criteria:

* TMJ deformity due to osteoarthrosis, ankylosis, injury, and pathology
* medicaly free patients

Exclusion Criteria:

* bilateral TMJ deformity
* patients medically compromised

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 2 weeks
  0 representing no pain and 10 representing the highest level of pain
inflammation score scale | 1 month
  0 no inflammation, 1-3 mild inflammation,4-7 moderate inflammation,8-10 severe inflammation

SECONDARY OUTCOMES:
mouth opening | 6 months
  normal ranged from 33 mm to 38 mm

CONTACTS AND LOCATIONS:
Overall Officials: Marwa T Ibrahim, Ass prof, Principal Investigator — Tanta University
Locations (1):
- Egypt, Tanta, Egypt